CLINICAL TRIAL: NCT02404220
Title: A Phase 1b/2, Open-Label, Dose Escalation and Expansion Study Evaluating the Safety and Efficacy of Entospletinib (GS-9973) With Vincristine and Dexamethasone in Adult Subjects With Relapsed or Refractory Acute Lymphoblastic Leukemia (ALL)
Brief Title: Safety and Efficacy of Entospletinib With Vincristine and Dexamethasone in Adults With Relapsed or Refractory Acute Lymphoblastic Leukemia (ALL)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-339-1560; 2015-002768-18 (EudraCT Number)
Record Dates: First submitted 2015-03-02; First posted 2015-03-31 (Estimated); Results first posted 2019-12-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Syk inhibitor; Blood malignancy; Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — 6-(1H-indazol-6-yl)-N-(4-morpholinophenyl)imidazo(1,2-a)pyrazin-8-amine; Vincristine; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ENTO 200 mg + VCR 0.5 mg (Experimental): Monotherapy Lead-In (Day -7 to Day -1): Entospletinib (ENTO) 200 mg tablet orally twice daily as a single agent.
  Induction (two 28-day cycles): ENTO 200 mg twice daily continuously in combination with vincristine (VCR) 0.5 mg intravenously (IV) on Days 1, 8, 15, and 22 of each cycle; dexamethasone (DEX) 20 mg twice daily orally on Days 8-11 and Days 22-25 (Cycle 1) and on Days 1-4 and Days 15-18 (Cycle 2); and central nervous system (CNS) prophylaxis per institutional standards on Day 28 of each cycle.
  Maintenance (up to 36, 28-day cycles): Participants who achieved a complete remission (CR) received stem cell transplant (SCT) (if eligible) per investigator's discretion; others who obtained clinical benefit (ie, at least a partial response [PR]) after induction were offered maintenance therapy with ENTO 200 mg twice daily continuously in combination with VCR 0.5 mg on Day 1 of each cycle and DEX (20 mg daily or 10 mg twice daily) on Days 1-4 and Days 15-18 of each cycle.
  Interventions: Drug: Entospletinib; Drug: Vincristine; Drug: Dexamethasone; Drug: CNS Prophylaxis
- ENTO 400 mg + VCR 0.5 mg (Experimental): Monotherapy Lead-In (Day -7 to Day -1): ENTO 400 mg tablet orally twice daily as a single agent.
  Induction (two 28-day cycles): ENTO 400 mg twice daily continuously in combination with VCR 0.5 mg IV on Days 1, 8, 15, and 22 of each cycle; DEX 20 mg twice daily orally on Days 8-11 and Days 22-25 (Cycle 1) and on Days 1-4 and Days 15-18 (Cycle 2); and CNS prophylaxis per institutional standards on Day 28 of each cycle.
  Maintenance (up to 36, 28-day cycles): Participants who achieved a CR received SCT (if eligible) per investigator's discretion; others who obtained clinical benefit (ie, at least a PR) after induction were offered maintenance therapy with ENTO 400 mg twice daily continuously in combination with VCR 0.5 mg on Day 1 of each cycle and DEX (20 mg daily or 10 mg twice daily) on Days 1-4 and Days 15-18 of each cycle.
  Interventions: Drug: Entospletinib; Drug: Vincristine; Drug: Dexamethasone; Drug: CNS Prophylaxis
- ENTO 400 mg + VCR 1.0 mg (Experimental): Monotherapy Lead-In (Day -7 to Day -1): ENTO 400 mg tablet orally twice daily as a single agent.
  Induction (two 28-day cycles): ENTO 400 mg twice daily continuously in combination with VCR 1.0 mg IV on Days 1, 8, 15, and 22 of each cycle; DEX 20 mg twice daily orally on Days 8-11 and Days 22-25 (Cycle 1) and on Days 1-4 and Days 15-18 (Cycle 2); and CNS prophylaxis per institutional standards on Day 28 of each cycle.
  Maintenance (up to 36, 28-day cycles): Participants who achieved a CR received SCT (if eligible) per investigator's discretion; others who obtained clinical benefit (ie, at least a PR) after induction were offered maintenance therapy with ENTO 400 mg twice daily continuously in combination with VCR 1.0 mg on Day 1 of each cycle and DEX (20 mg daily or 10 mg twice daily) on Days 1-4 and Days 15-18 of each cycle.
  Interventions: Drug: Entospletinib; Drug: Vincristine; Drug: Dexamethasone; Drug: CNS Prophylaxis
- ENTO 400 mg + VCR 2.0 mg (Experimental): Monotherapy Lead-In (Day -7 to Day -1): ENTO 400 mg tablet orally twice daily as a single agent.
  Induction (two 28-day cycles): ENTO 400 mg twice daily continuously in combination with VCR 2.0 mg IV on Days 1, 8, 15, and 22 of each cycle; DEX 20 mg twice daily orally on Days 8-11 and Days 22-25 (Cycle 1) and on Days 1-4 and Days 15-18 (Cycle 2); and CNS prophylaxis per institutional standards on Day 28 of each cycle.
  Maintenance (up to 36, 28-day cycles): Participants who achieved a CR received SCT (if eligible) per investigator's discretion; others who obtained clinical benefit (ie, at least a PR) after induction were offered maintenance therapy with ENTO 400 mg twice daily continuously in combination with VCR 2.0 mg on Day 1 of each cycle and DEX (20 mg daily or 10 mg twice daily) on Days 1-4 and Days 15-18 of each cycle.
  Interventions: Drug: Entospletinib; Drug: Vincristine; Drug: Dexamethasone; Drug: CNS Prophylaxis

INTERVENTIONS:
Drug: Entospletinib
  Other Names: GS-9973; ENTO
Drug: Vincristine
  Other Names: VCR
Drug: Dexamethasone
  Other Names: DEX
Drug: CNS Prophylaxis

SUMMARY:
The primary objective of this study is to evaluate the safety of entospletinib in combination with vincristine (VCR), and dexamethasone (DEX) in adults with previously treated relapsed or refractory B-cell lineage acute lymphoblastic leukemia (ALL).

This is a dose escalation study in which after 2 induction cycles participants may be put on maintenance for up to 36 cycles if they have obtained clinical benefit from the treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Adults with ALL in need of treatment

Key Exclusion Criteria:

* Diagnosis of Burkitt's Leukemia, or lymphoid blast crisis of chronic myelogenous leukemia (CML)
* History of myelodysplastic syndrome or solid organ transplantation
* Prior allogeneic bone marrow progenitor cell transplant within 100 days or on active immunosuppression for graft versus host disease (GVHD) treatment or prophylaxis within 28 days prior to enrollment

Note: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-05-06 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (13):
- United States (10):
  - City of Hope, Duarte, California
  - UCLA, Los Angeles, California
  - UC Irvine Medical Center, Orange, California
  - University of California San Diego (UCSD), San Diego, California
  - University of Chicago, Chicago, Illinois
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan-Kettering, New York, New York
  - The Ohio State University, Columbus, Ohio
  - Bon Secour St. Francis Hospital, Greenville, South Carolina
  - University of WA, Seattle, Washington
- Princess Margaret, Toronto, Ontario, Canada
- Germany (2):
  - Medizinische Klinik mit Schwerpunkt Hepatologie & Gastroenterology, Berlin
  - Medizinische Klinik und Poliklinik I, Würzburg

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Germany, Canada, and United States. The first participant was screened on 06 May 2015. The last study visit occurred on 17 December 2018.
Pre-assignment Details: 42 participants were screened.
Period: Overall Study
Arm/Group | ENTO 200 mg + VCR 0.5 mg | ENTO 400 mg + VCR 0.5 mg | ENTO 400 mg + VCR 1.0 mg | ENTO 400 mg + VCR 2.0 mg
Started | 5 | 8 | 7 | 10
Completed | 0 | 0 | 0 | 0
Not Completed | 5 | 8 | 7 | 10
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Death | 5 | 5 | 3 | 8
Not completed — Progressive Disease | 0 | 0 | 1 | 1
Not completed — Study Terminated by Sponsor | 0 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Enrolled but Never Treated | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Enrolled Analysis Set included all participants who received a study identification number in the study after screening.
Groups:
- ENTO 200 mg + VCR 0.5 mg: Monotherapy Lead-In (Day -7 to Day -1): ENTO 200 mg tablet orally twice daily as a single agent.
  Induction (two 28-day cycles): ENTO 200 mg twice daily continuously in combination with VCR 0.5 mg IV on Days 1, 8, 15, and 22 of each cycle; DEX 20 mg twice daily orally on Days 8-11 and Days 22-25 (Cycle 1) and on Days 1-4 and Days 15-18 (Cycle 2); and CNS prophylaxis per institutional standards on Day 28 of each cycle.
  Maintenance (up to 36, 28-day cycles): Participants who achieved a CR received SCT (if eligible) per investigator's discretion; others who obtained clinical benefit (ie, at least a PR) after induction were offered maintenance therapy with ENTO 200 mg twice daily continuously in combination with VCR 0.5 mg on Day 1 of each cycle and DEX (20 mg daily or 10 mg twice daily) on Days 1-4 and Days 15-18 of each cycle.
- Total: Total of all reporting groups
Arm/Group | ENTO 200 mg + VCR 0.5 mg | ENTO 400 mg + VCR 0.5 mg | ENTO 400 mg + VCR 1.0 mg | ENTO 400 mg + VCR 2.0 mg | Total
Number analyzed (Participants) | 5 | 8 | 7 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Participants in Full Analysis Set (all participants who received at least 1 dose of study treatment) were analyzed.
  years
    number analyzed (Participants) | 5 | 6 | 7 | 10 | 28
    (all) | 46.8 (16.93) | 51.7 (17.72) | 47.4 (9.68) | 52.7 (19.66) | 50.1 (16.04)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participants in Full Analysis Set were analyzed.
  Participants
    number analyzed (Participants) | 5 | 6 | 7 | 10 | 28
    Female | 5 | 4 | 2 | 3 | 14
    Male | 0 | 2 | 5 | 7 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Participants in Full Analysis Set were analyzed.
  Participants
    Race: number analyzed (Participants) | 5 | 6 | 7 | 10 | 28
    Race: Asian | 1 | 0 | 1 | 0 | 2
    Race: Black | 0 | 0 | 1 | 0 | 1
    Race: White | 4 | 5 | 5 | 10 | 24
    Race: Not Permitted | 0 | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Participants in Full Analysis Set were analyzed.
  Participants
    Ethnicity: number analyzed (Participants) | 5 | 6 | 7 | 10 | 28
    Ethnicity: Hispanic or Latino | 1 | 2 | 2 | 5 | 10
    Ethnicity: Not Hispanic or Latino | 4 | 3 | 5 | 5 | 17
    Ethnicity: Not Permitted | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 0 | 1 | 0 | 0 | 1
  United States | 5 | 7 | 6 | 9 | 27
  Germany | 0 | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Dose Limiting Toxicities (DLTs)
Description: The occurrence of any of the following toxicities during Lead-in/Cycle 1 (Day -7 through Day 28) was considered a DLT if judged by the investigator to be possibly, probably, or definitely related to the administration of any drug in the treatment regimen (ENTO, VCR, DEX, institutional standard CNS prophylaxis):
  * Grade 4 (or higher) non-hematologic toxicity
  * Grade 3 non-hematologic toxicity lasting ≥ 7 days despite optimal supportive care
  * Any Grade 3 non-hematologic laboratory value if:
    * Medical intervention was required to treat, or
    * The abnormality led to hospitalization, or
    * The abnormality persisted for > 1 week
  * Grade 4 Neutropenia (absolute neutrophil count [ANC] < 500 /μL) persistent for greater than 14 days or associated with febrile neutropenia
  * Grade 4 thrombocytopenia (platelets < 25,000/μL) persisting for greater than 14 days (or greater than 25,000 /μL, but requiring prophylactic platelet transfusion to maintain this level)
Time Frame: ENTO Lead-in and Cycle 1 (Day -7 through Day 28)
Population: DLT Analysis Set included all participant in the Safety Analysis Set (all participants who received at least 1 dose of study treatment) who met at least one of the following criteria: received at least 21 days of ENTO, > 50% of planned total dose of VCR and DEX, or experienced a DLT during the DLT assessment window.
Measure: Number; unit: percentage of participants
Arm/Group | ENTO 200 mg + VCR 0.5 mg | ENTO 400 mg + VCR 0.5 mg | ENTO 400 mg + VCR 1.0 mg | ENTO 400 mg + VCR 2.0 mg
Number analyzed (Participants) | 3 | 3 | 6 | 7
percentage of participants | 33.3 | 0 | 16.7 | 0

2. Secondary Outcome: Percentage of Participants With Complete Remission (CR) at the End of Induction
Description: Assessment of clinical response was made according to National Comprehensive Cancer Network (NCCN) guidelines on acute lymphoblastic leukemia (ALL) Version 2, 2016. CR required all of the following:
  * No circulating blasts or extramedullary disease (no lymphadenopathy, splenomegaly, skin/gum infiltration/testicular mass/CNS involvement).
  * Trilineage hematopoiesis (TLH) and < 5% blasts in bone marrow aspirate.
  * ANC > 1000/μL.
  * Platelets > 100,000/μL.
Time Frame: End of Induction (Cycle 2, Day 28)
Population: The Full Analysis Set included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | ENTO 200 mg + VCR 0.5 mg | ENTO 400 mg + VCR 0.5 mg | ENTO 400 mg + VCR 1.0 mg | ENTO 400 mg + VCR 2.0 mg
Number analyzed (Participants) | 5 | 6 | 7 | 10
percentage of participants | 20.0 | 33.3 | 14.3 | 0

3. Secondary Outcome: Percentage of Participants With Overall Remission at the End of Induction
Description: Assessment of clinical response was made according to NCCN guidelines on ALL Version 2, 2016. Overall remission included CR and complete remission with incomplete hematologic recovery (CRi). CR required all of the following:
  * No circulating blasts or extramedullary disease (no lymphadenopathy, splenomegaly, skin/gum infiltration/testicular mass/CNS involvement).
  * TLH and < 5% blasts in bone marrow aspirate.
  * ANC > 1000/μL.
  * Platelets > 100,000/μL.
  CRi required all criteria for CR except platelet count and/or ANC:
  * Platelets ≤ 100,000/μL and/or ANC is ≤ 1000/μL
Time Frame: End of Induction (Cycle 2, Day 28)
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | ENTO 200 mg + VCR 0.5 mg | ENTO 400 mg + VCR 0.5 mg | ENTO 400 mg + VCR 1.0 mg | ENTO 400 mg + VCR 2.0 mg
Number analyzed (Participants) | 5 | 6 | 7 | 10
percentage of participants | 20.0 | 33.3 | 14.3 | 0.0

4. Secondary Outcome: Percentage of Participants With Partial Response (PR) at the End of Induction
Description: PR required all of the following:
  * No circulating blasts or extramedullary disease (no lymphadenopathy, splenomegaly, skin/gum infiltration/testicular mass/CNS involvement).
  * TLH and bone marrow may contain ≥ 5% but less than 25% blast morphology.
  * ANC > 1000/μL.
  * Platelets > 100,000/μL.
Time Frame: End of Induction (Cycle 2, Day 28)
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | ENTO 200 mg + VCR 0.5 mg | ENTO 400 mg + VCR 0.5 mg | ENTO 400 mg + VCR 1.0 mg | ENTO 400 mg + VCR 2.0 mg
Number analyzed (Participants) | 5 | 6 | 7 | 10
percentage of participants | 0.0 | 0.0 | 14.3 | 10.0

5. Secondary Outcome: Percentage of Participants With Overall Response at the End of Induction
Description: Overall response included CR, CRi, and PR. CR required all of the following:
  * No circulating blasts or extramedullary disease (no lymphadenopathy, splenomegaly, skin/gum infiltration/testicular mass/CNS involvement).
  * TLH and < 5% blasts in bone marrow aspirate.
  * ANC > 1000/μL.
  * Platelets > 100,000/μL.
  CRi required all criteria for CR except platelet count and/or ANC:
  * Platelets ≤ 100,000/μL and/or ANC is ≤ 1000/μL
  PR required all criteria for CR except for bone marrow blasts:
  * bone marrow may contain ≥ 5% but less than 25% blast morphology
Time Frame: End of Induction (Cycle 2, Day 28)
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | ENTO 200 mg + VCR 0.5 mg | ENTO 400 mg + VCR 0.5 mg | ENTO 400 mg + VCR 1.0 mg | ENTO 400 mg + VCR 2.0 mg
Number analyzed (Participants) | 5 | 6 | 7 | 10
percentage of participants | 20.0 | 33.3 | 28.6 | 10.0

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to maximum 18 months; All-Cause Mortality: First dose date up to maximum 3.5 years
Description: The Safety Analysis Set included all participants who received at least 1 dose of study treatment.
Arm/Group | ENTO 200 mg + VCR 0.5 mg | ENTO 400 mg + VCR 0.5 mg | ENTO 400 mg + VCR 1.0 mg | ENTO 400 mg + VCR 2.0 mg
All-Cause Mortality (participants affected / at risk) | 5/5 | 5/6 | 5/7 | 9/10
Serious Adverse Events (participants affected / at risk) | 5/5 | 4/6 | 5/7 | 6/10
Other Adverse Events (participants affected / at risk) | 5/5 | 5/6 | 6/7 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ENTO 200 mg + VCR 0.5 mg (N=5) | ENTO 400 mg + VCR 0.5 mg (N=6) | ENTO 400 mg + VCR 1.0 mg (N=7) | ENTO 400 mg + VCR 2.0 mg (N=10)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 1 | 0
Fungaemia (Infections and infestations) | 1 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 2 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis fungal (Infections and infestations) | 1 | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ENTO 200 mg + VCR 0.5 mg (N=5) | ENTO 400 mg + VCR 0.5 mg (N=6) | ENTO 400 mg + VCR 1.0 mg (N=7) | ENTO 400 mg + VCR 2.0 mg (N=10)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 0
Haemolysis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 2 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Cushingoid (Endocrine disorders) | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0
Eye haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 4 | 4 | 2
Oral disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1
Catheter site erythema (General disorders) | 0 | 1 | 0 | 0
Catheter site haemorrhage (General disorders) | 1 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 1
Chills (General disorders) | 1 | 0 | 1 | 0
Crepitations (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 3 | 2 | 2 | 3
Feeling cold (General disorders) | 1 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 1 | 1
Malaise (General disorders) | 0 | 0 | 2 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 2 | 2 | 0 | 1
Pain (General disorders) | 0 | 1 | 0 | 0
Puncture site pain (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 3 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis fungal (Infections and infestations) | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 1 | 2
Blood bilirubin increased (Investigations) | 2 | 1 | 0 | 0
Blood immunoglobulin G decreased (Investigations) | 1 | 0 | 0 | 0
Escherichia test positive (Investigations) | 1 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 1 | 1 | 1 | 3
Platelet count decreased (Investigations) | 0 | 1 | 2 | 2
Staphylococcus test positive (Investigations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 1 | 0 | 3
White blood cell count increased (Investigations) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0 | 1 | 2
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 1 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 2 | 2
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 1 | 1 | 1
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 3 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Device malfunction (Product Issues) | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0
Fear (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 2 | 4
Irritability (Psychiatric disorders) | 0 | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1 | 1
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 2 | 0
Hypotension (Vascular disorders) | 1 | 1 | 1 | 0
Pallor (Vascular disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to the low response rate observed with ENTO + VCR + DEX in adults with relapsed or refractory B-ALL, the sponsor decided not to proceed with Phase 2 (dose-expansion) and the cohort was subsequently closed with no participant enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-12-03): https://cdn.clinicaltrials.gov/large-docs/20/NCT02404220/SAP_000.pdf
  • Study Protocol: Amendment 5 (2018-04-13): https://cdn.clinicaltrials.gov/large-docs/20/NCT02404220/Prot_001.pdf